CLINICAL TRIAL: NCT05612555
Title: Low Psoas Index and Cardiac Assistance: No Excess Mortality at D28 Post Implantation
Acronym: VAD
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7531
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Ventricular Assist Device
Keywords: Ventricular Assist Device; VAD; Sarcopenia; Psoas Index; Cardiac assistance; Cardiac assistance surgery
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The frailty syndrome is important to consider in perioperative cardiac assistance. One of its components is the patient's sarcopenia. This can be assessed by measuring the size of the psoas muscle. For this purpose, one of the most studied measures seems to be the measurement of the Psoas Index. This is a contouring of the psoas muscle, performed on an axial section of a CT scan, at the level of the L4 vertebra, which is then matched to the body surface. However, there is no standardization of measurements and volume acquisitions, and different image processing is also described. A radiological evaluation of the psoas could overcome this difficulty and provide a rapid and available screening tool for sarcopenia.

ELIGIBILITY:
Inclusion criteria:

* Major subject ((≥18 years old)
* Subject who underwent surgery for placement of a ventricular assist device between 01/02/2014 and 30/06/2018
* Subject who has not expressed opposition to the reuse of his or her data for research purposes

Exclusion Criteria:

* Subject having expressed opposition to participate in the study
* Absence of CT scan available at the time of implantation or CT scans older than one year prior to surgery and those older than 72 hours postoperatively
* No anthropometric data available
* Subject under legal protection
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject ((≥18 years old) having surgery for placement of a ventricular assist device between 01/02/2014 and 30/06/2018 in Strasbourg University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Impact of sarcopenia, measured by the Psoas Index, on 28-day survival in patients undergoing cardiac assistance surgery | Survival at 28 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Réanimation Chirurgicale - CHU de Strasbourg - France, Strasbourg, France